CLINICAL TRIAL: NCT06424678
Title: Study of Cardiorespiratory Arrests That Occurred in the Surgical Block and Adjacent
Brief Title: Study of Cardiorespiratory Arrests That Occurred in the Surgical Block and Adjacent Places
Status: Not yet recruiting | Type: Observational
Sponsor: Sociedad Española de Anestesiología, Reanimación y Terapéutica del Dolor (Other)
Responsible Party: Principal Investigator, Maria Concepcion Ruiz-Villen, Doctor (PhD) in Medicine and Surgery. Faculty specialist in Anaesthesiology, Intensive Care and Pain, Sociedad Española de Anestesiología, Reanimación y Terapéutica del Dolor
Other Study IDs: SeRCP022024
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Cardiorespiratory Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cradiorespiratory arrest in paediatric patients: The epidemiology of the data collected in the Utstein template will be described in patients who suffer cardiac arrest in the surgical block and have an age between 1 month and 1 day to 18 years.
  Interventions: Other: Only data collection in the Utstein template
- cardiorespiratory arrest in adult patients: The epidemiology of the data collected in the Utstein template will be described in patients who suffer cardiac arrest in the surgical block and are aged from 18 years and 1 day to 11o years.
  Interventions: Other: Only data collection in the Utstein template

INTERVENTIONS:
Other: Only data collection in the Utstein template — The intervention that we will carry out in both groups will consist of collecting data from the patient (age, sex and race), on cardiopulmonary arrest, cardiopulmonary resuscitation, and the results of cardiopulmonary resuscitation.

SUMMARY:
A protocol for recording cardiopulmonary arrest (CRP) data in the in-hospital surgical block has been designed with the Utstein template model. The database is hosted in accordance with European legislation on patient data protection.

Invitation to participate will be sent to Spanish hospitals in the first phase. Once this is over, participation in the registry will be opened to European hospitals. Survival and neurological outcome will be evaluated upon discharge from the surgical block. The study design is a prospective observational registry of a cohort of subjects who have suffered a CRP in the surgical block.

DETAILED DESCRIPTION:
Patients will be enrolled by participating researchers from Spanish hospitals that have a pediatric surgery service, in addition to surgery on adult patients, who will collect and upload the data into a protected web-based electronic database. The recorded variables are grouped as follows: patient variables, hospital data, data prior to cardiopulmonary arrest (CRP), data from cardiopulmonary arrest (CRP), data after cardiopulmonary resuscitation (CPR), results of cardiopulmonary resuscitation (CPR). For the study, cardiorespiratory arrest (CRP) is defined as cardiac arrest for which resuscitation is attempted with chest compressions, defibrillation, or both. In the pediatric population it may include patients receiving chest compressions for poor perfusion in the setting of severe bradycardia.

The inclusion criteria are: all patients older than 1 month who undergo sedation, anesthesia or monitored anesthetic surveillance performed by an anesthesiologist and suffer cardiorespiratory arrest in the surgical block. Subsequent episodes of cardiorespiratory arrest (CRP) in the same subject may be included. Exclusion criteria: hospitals that do not have a pediatric surgery service in their service portfolio, patients being treated with extracorporeal circulatory support (ECMO, extracorporeal circulation pump or ventricular assistance) at the time of cardiorespiratory arrest. Patients who suffer cardiac arrest and require any type of extracorporeal circulatory support for the recovery of spontaneous circulation after performing the corresponding cardiopulmonary resuscitation (CPR) will not be eliminated.

The data collection period will be valid for 48 months, starting on June 1, 2025 and the last day being June 1, 2029.

ELIGIBILITY:
Inclusion Criteria:Patients over 1 month of age who suffer cardiac arrest in the surgical unit and/or in those places where some type of monitored surveillance technique, sedation and/or anesthesia is performed by an anesthesiologist or internal resident specialist (EIR) of the specialty of Anesthesiology.

Exclusion Criteria:

* Patients with procedures defined as major outpatient surgery in the hospital where the cardiac arrest occurs.
* Patients in supportive treatment extracorporeal circulatory system (ECMO) or ventricular assist at the time of cardiac arrest.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients over 1 month of age who suffer cardiac arrest in the surgical block (BQ). Cardiac arrest is defined by the application of chest compressions and/or defibrillation. In the pediatric population it may include patients receiving chest compressions for poor perfusion in the setting of severe bradycardia.
  We define BQ as "the space in which all the operating rooms are grouped, with the equipment and characteristics necessary to carry out all the planned surgical procedures. The BQ includes the premises where the care process of the surgical procedure takes place (operating room and post-anesthesia recovery unit) and the support premises it requires. In these locations we include the pre-operating room where patients wait, within the surgical block, to enter the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Survival to discharge from the surgical block will be evaluated | From June 1, 2025 to June 1, 2029
  We define survival upon discharge from the BQ as that patient with recovery of spontaneous circulation after cardiac arrest, who is discharged with signs of life to the hospital ward.

SECONDARY OUTCOMES:
Survival to hospital discharge with good neurological status | From June 1, 2025 to June 1, 2029
  Neurological outcome at 30 days or at hospital discharge if it occurs before that period. Registers as Cerebral Performance Category (CPC), Pediatric CPC (PCPC), or modified Rankin Scale (mRS) score, and can be measured face-to-face, telephone interview, or a combination. The PCC is a 5-point scale ranging from 1 (good brain performance) to 5 (dead). The PCPC is a scale that goes from 1 (good brain performance) to 6 (dead). The mRS is a scale that ranges from 0 (no symptoms) to 6 (dead). Survival with favorable neurological conditions is defined as a CPC of 1 or 2, mRS of 0 to 3, or no change in CPC or mRS with respect to the patient's pre-arrest status. Include a definition of how it was measured (face- to-face, extracted from notes, combination.

CONTACTS AND LOCATIONS:
Overall Officials: María Conepción Ruiz-Villén, Principal Investigator — Sociedad Española de Anestesiología, Reanimación y Terapéutica del Dolor

IPD SHARING:
Plan to Share IPD: Undecided
Data collected in the Utstein template can be shared with other SEDAR researchers. The data will be encrypted.

REFERENCES:
- [Background] Berg KM, Bray JE, Ng KC, Liley HG, Greif R, Carlson JN, Morley PT, Drennan IR, Smyth M, Scholefield BR, Weiner GM, Cheng A, Djarv T, Abelairas-Gomez C, Acworth J, Andersen LW, Atkins DL, Berry DC, Bhanji F, Bierens J, Bittencourt Couto T, Borra V, Bottiger BW, Bradley RN, Breckwoldt J, Cassan P, Chang WT, Charlton NP, Chung SP, Considine J, Costa-Nobre DT, Couper K, Dainty KN, Dassanayake V, Davis PG, Dawson JA, Fernanda de Almeida M, De Caen AR, Deakin CD, Dicker B, Douma MJ, Eastwood K, El-Naggar W, Fabres JG, Fawke J, Fijacko N, Finn JC, Flores GE, Foglia EE, Folke F, Gilfoyle E, Goolsby CA, Granfeldt A, Guerguerian AM, Guinsburg R, Hatanaka T, Hirsch KG, Holmberg MJ, Hosono S, Hsieh MJ, Hsu CH, Ikeyama T, Isayama T, Johnson NJ, Kapadia VS, Daripa Kawakami M, Kim HS, Kleinman ME, Kloeck DA, Kudenchuk P, Kule A, Kurosawa H, Lagina AT, Lauridsen KG, Lavonas EJ, Lee HC, Lin Y, Lockey AS, Macneil F, Maconochie IK, John Madar R, Malta Hansen C, Masterson S, Matsuyama T, McKinlay CJD, Meyran D, Monnelly V, Nadkarni V, Nakwa FL, Nation KJ, Nehme Z, Nemeth M, Neumar RW, Nicholson T, Nikolaou N, Nishiyama C, Norii T, Nuthall GA, Ohshimo S, Olasveengen TM, Gene Ong YK, Orkin AM, Parr MJ, Patocka C, Perkins GD, Perlman JM, Rabi Y, Raitt J, Ramachandran S, Ramaswamy VV, Raymond TT, Reis AG, Reynolds JC, Ristagno G, Rodriguez-Nunez A, Roehr CC, Rudiger M, Sakamoto T, Sandroni C, Sawyer TL, Schexnayder SM, Schmolzer GM, Schnaubelt S, Semeraro F, Singletary EM, Skrifvars MB, Smith CM, Soar J, Stassen W, Sugiura T, Tijssen JA, Topjian AA, Trevisanuto D, Vaillancourt C, Wyckoff MH, Wyllie JP, Yang CW, Yeung J, Zelop CM, Zideman DA, Nolan JP; ; and Collaborators. 2023 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations: Summary From the Basic Life Support; Advanced Life Support; Pediatric Life Support; Neonatal Life Support; Education, Implementation, and Teams; and First Aid Task Forces. Resuscitation. 2024 Feb;195:109992. doi: 10.1016/j.resuscitation.2023.109992. Epub 2023 Nov 9. PMID 37937881
- [Background] Nolan JP, Berg RA, Andersen LW, Bhanji F, Chan PS, Donnino MW, Lim SH, Ma MH, Nadkarni VM, Starks MA, Perkins GD, Morley PT, Soar J. Cardiac Arrest and Cardiopulmonary Resuscitation Outcome Reports: Update of the Utstein Resuscitation Registry Template for In-Hospital Cardiac Arrest: A Consensus Report From a Task Force of the International Liaison Committee on Resuscitation (American Heart Association, European Resuscitation Council, Australian and New Zealand Council on Resuscitation, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Southern Africa, Resuscitation Council of Asia). Circulation. 2019 Oct 29;140(18):e746-e757. doi: 10.1161/CIR.0000000000000710. Epub 2019 Sep 16. PMID 31522544
- [Background] Ministerio de Sanidad y política social.Bloque Quirúrgico. Estándares y recomendaciones. Madrid. Centro de publicaciones. 2009.301 p.